CLINICAL TRIAL: NCT07320794
Title: The Effect of Mindfulness Training on Coping With Fear of Birth Training Applied Online to Pregnant Women on Fear of Birth and Birth Satisfaction
Brief Title: The Effect of Mindful Awareness on Fear and Satisfaction of Childbirth.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Funda ÇINAR SAY, Principal Investigator, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: Interventional(clinical) Trial
Record Dates: First submitted 2025-12-22; First posted 2026-01-06 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Fear of Childbirth; Mindfulness
Keywords: Mindfulness; Fear of childbirth; Birth satisfaction; Midwifery, Education

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral: Intervention group (Experimental): The mindfulness training was conducted over three weeks, with two sessions per week, for a total of six sessions. Pregnant women were given brochures and booklets prepared by the researcher, appropriate to the training content, before the training (Appendix 13). Pregnant women in the intervention group received training reminders via text message the day before the training and again via text message a few hours before the training, sometimes by phone. The training was conducted at times convenient for the pregnant women, with each session lasting 40-45 minutes. At least two weeks after the mindfulness training, data were collected online using the W-DEQ-A and mindfulness scales; those who could not be reached were administered face-to-face, and those who could not be reached were administered via text message. Between days 7 and 15 postpartum, the postpartum information form, the W-DEQ-B and mindfulness scales, and the birth satisfaction scale were administered to the women at times
  Interventions: Behavioral: Mindfulness-Based Childbirth Education
- control group (No Intervention): No Intervention: Control group The control group continued to receive the routine care

INTERVENTIONS:
Behavioral: Mindfulness-Based Childbirth Education — The intervention consisted of a structured mindfulness-based childbirth education program delivered over three weeks, with two sessions per week (six sessions in total). Each session lasted approximately 40-45 minutes. The program aimed to reduce fear of childbirth and improve childbirth satisfaction. Educational materials were provided to participants, and reminder messages were sent before each session.
  Other Names: Intervention group
  Arms: Behavioral: Intervention group

SUMMARY:
The aim of this study is to conduct a randomized controlled experimental study to determine the effect of online mindfulness-based childbirth anxiety training on childbirth anxiety and birth satisfaction in pregnant women.

DETAILED DESCRIPTION:
The aim of this study is to conduct a randomized controlled experimental study to determine the effect of online mindfulness-based childbirth anxiety training on childbirth anxiety and birth satisfaction in pregnant women.

Detailed Description: Childbirth anxiety is a common problem among women and affects their health and well-being before, during, and after pregnancy.

This problem can lead to negative pregnancy outcomes and can also cause psychological problems for the woman.

Childbirth anxiety can also affect the choice of delivery method and lead to an increase in cesarean section rates.

Healthcare services provided by midwives and other healthcare professionals during pregnancy and childbirth have the power to reduce or increase childbirth anxiety.

The most important midwifery intervention that can be used to reduce childbirth anxiety is counseling. The importance of childbirth anxiety for the midwifery profession is clearly evident from the fact that women prefer more interventions during childbirth. Large epidemiological studies provide good evidence that women experiencing childbirth anxiety prefer interventions during childbirth. When mindfulness training is examined in general, it is seen that mindfulness-based interventions can be effective in increasing positive emotions and decreasing negative emotions. The use of mindfulness-based interventions is increasing day by day, and their clinical benefits are being proven by studies. In light of these studies, it can be said that the method can be used in women not only to reduce stress but also as an effective method with physiological benefits. It is necessary to increase basic mindfulness training for pregnant women, to include midwives in mindfulness-based interventions, to develop intervention programs for women's specific life stages by ensuring necessary collaborations, and to evaluate the results of these programs. Studies have indicated that mindfulness training during counseling increases women's self-esteem. With mindfulness training, pregnant women's sense of control and self-confidence during childbirth can be increased, and birth outcomes can be improved positively. This study was conducted to determine the effect of mindfulness-based childbirth fear management training given to women on childbirth fear and birth satisfaction. The hypothesis that there was no difference in the mean childbirth fear and satisfaction scores between the intervention and control groups after the intervention was tested.

ELIGIBILITY:
Inclusion Criteria:

* Between 20-35 years of age,
* At least a secondary school graduate,
* Residing within the borders of Aydın province,
* Being between 28-32 weeks pregnant according to the last menstrual period,
* Having no obstacles to giving birth vaginally,
* Having decided to give birth vaginally,
* Having the conditions to receive online training (internet, computer, smartphone, etc.),
* Being able to speak and understand Turkish,
* Pregnant women who are having their first pregnancy will be included.

Exclusion Criteria:

* • Women whose current pregnancy is high-risk (such as multiple pregnancy, preeclampsia, diabetes, heart disease, placenta previa, oligohydramnios),

  * Women diagnosed with mental illnesses (depression, anxiety disorder, schizophrenia, bipolar disorder, etc.),
  * All pregnant women who have undergone infertility treatment and become pregnant will not be included in the study.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2025-01-06 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
2. Fear of childbirth after intervention | [Time Frame: 37-40 gestational weeks]
  2. Fear of childbirth after intervention assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version A. This instrument contains questions on women's prenatal expectations to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel before their delivery. This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version A is based on a 6-point Likert scale numbered 0-5. Zero corresponds to the response, "Totally" and five means "none." The minimum possible score on the scale is a "0"; maximum is 165. Higher scores indicate greater levels of Fear of Childbirth. [Time Frame: 36-38 gestational weeks]
Fear of childbirth before intervention | [Time Frame: 28-32 gestational weeks
  . Fear of childbirth before intervention assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version A. This instrument contains questions on women's prenatal expectations to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel before their delivery. This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version A is based on a 6-point Likert scale numbered 0-5. Zero corresponds to the response, "Totally" and five means "none." The minimum possible score on the scale is a "0"; maximum is 165. Higher scores indicate greater levels of Fear of Childbirth.
Fear of childbirth after birth | [Time Frame: 7-15 day after the birth]
  Fear of childbirth after birth assessed using the Wijma Delivery Expectancy/Experience Questionnaire- Version B. This instrument contains questions on women's postpartum experiences to measure the nature of the fear experienced during and following childbirth. The instrument makes it possible to identify the nature of the fear of childbirth women feel after their delivery.
  This scale contain 33 questions. Wijma Delivery Expectancy/Experience Questionnaire- Version-B is based on a 6- point Likert scale where the responses are numbered from 1-6 and one corresponds to the response, "Totally" and six means "none." The total possible score on the scale varies between 33-198. Higher scores indicate greater levels of Fear of Childbirth.
Birth satisfaction scale. | [Time Frame: 7-15 days after birth
  Birth satisfaction scale. Each item is rated on a four-point Likert scale (1=strongly agree, 2=partially agree, 3=somewhat agree, 4=strongly disagree). A minimum score of 10 and a maximum score of 40 are accepted. There is no cutoff point on the scale. A high score is associated with low birth satisfaction.
  [Time Frame: 7-15 days after birth]

SECONDARY OUTCOMES:
The Mindfulness Scale | Time Frame: 28-32 gestational weeks Time Frame: 37-40 gestational weeks Time Frame: 7-15. day after birth
  The Mindfulness Scale is a 15-item scale that measures the general tendency to be aware of and attentive to present experiences in daily life. The scale has a single-factor structure and gives a single total score. Higher scores on the scale indicate higher mindfulness. The scale is a 6-point Likert-type scale (Almost always, most of the time, sometimes, rarely, quite rarely, almost never).

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Aydin Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery, Aydin, Aydın
  - Aydin Adnan Menderes University, Faculty of Health Sciences, Division of Midwifery, Aydin

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: 6 months after publication
Access Criteria: elevance to the topic of the study and approval of all co-authors within 1 month of receiving the request.

REFERENCES:
- [Background] https://earsiv.odu.edu.tr/jspui/bitstream/11489/3915/1/10435776.pdf
- See also: Related Info — https://earsiv.odu.edu.tr/jspui/bitstream/11489/3915/1/10435776.pdf
- Available data/document: Clinical Study Report: fundacnr20@gmail.com — https://earsiv.odu.edu.tr/jspui/bitstream/11489/3915/1/10435776.pdf — https://earsiv.odu.edu.tr/jspui/bitstream/11489/3915/1/10435776.pdf
- Available data/document: Clinical Study Report: https://earsiv.odu.edu.tr/jspu — https://earsiv.odu.edu.tr/jspui/bitstream/11489/3915/1/10435776.pdf